CLINICAL TRIAL: NCT05352087
Title: Effect Of Early Versus Delayed Laparoscopic Cholecystectomy On Postoperative Mortality, Morbidity and Difficult Cholecystectomy In Patients With Grade II Cholecystitis According To Tokyo 2018 Guidelines: Prospective Randomised Study
Brief Title: Effect Of Early Versus Delayed Laparoscopic Cholecystectomy In Patients With Grade II Cholecystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gizem Kilinc Tuncer, General Surgery Consultant, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/134
Record Dates: First submitted 2022-04-19; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cholecystitis
Keywords: Acute cholecystitis; Laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early cholecystectomy (Active Comparator): In early cholecystectomy group after antibiotherapy was started with ceftriaxone and metronidazole, laparoscopic cholecystectomy was performed in the first 7 days following the hospitalization.
  Interventions: Procedure: Laparoscopic cholecystectomy
- delayed cholecystectomy (Active Comparator): Patients who accepted delayed surgery were also given the same antibiotherapy and operated after 6 weeks following their discharge
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is minimally invasive surgery to remove the gallbladder.

SUMMARY:
The timing ofthe cholecystectomy in patients with acute cholecystitis is still controversial. In our study, we aimed toinvestigate the effect of early and delayed cholecystectomy on difficultcholecystectomy, morbidity and mortality in patients diagnosed with Grade IIcholecystitis according to Tokyo 2018 guidelines.

DETAILED DESCRIPTION:
The timing ofthe cholecystectomy in patients with acute cholecystitis is still controversial. In our study, we aimed toinvestigate the effect of early and delayed cholecystectomy on difficultcholecystectomy, morbidity and mortality in patients diagnosed with Grade II cholecystitis according to Tokyo 2018 guidelines.

Patients that applied to the emergency department and diagnosed with Grade II acute cholecystitis between December 2019 and June 2021 were included in this study. Cholecystectomy was performed within 7 days and 6 weeks after symptom onset. The effect of early and delayed cholecystectomy was observed. The study is single-centered and the patient group graded as Grade II according to the Tokyo 2018 guideline acute cholecystitis diagnostic criteria will be included in the study. Patients will decide on the treatment method to be applied with their consent. The patients will be divided into two groups as those operated in the early period (first 7 days) and those operated in the late period (>6 weeks). The parameters to be compared were the rate of conversion from laparoscopic to open, bile duct injury and bile leakage rate, grade II-III complication rate in the Clavien Dindo complication scoring system, morbidity rate in the first 30 days postoperatively, and difficult cholecystectomy rate based on intraoperative imaging findings according to the Parkland scoring system. The research will be terminated when the number of 120 patients determined by the power analysis result is reached.

Chi-square and Student's t test will be used for the statistical evaluation of the results of the patients, respectively, for quantitative and continuous variables, and Mann-Whitney U test (two samples) or Kruskal-Wallis test (more than two samples) will be used for the analysis of abnormally distributed variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Grade II cholecystitis according to Tokyo 2018 guidelines
* Patients older than 18 years of age

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients diagnosed with choledocholithiasis
* Patients with Grade I or Grade III cholecystitis
* Pregnancy
* Patients unable to comply with the treatment or who could not consent to the treatment due to their mental state
* Patients that refused the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
mortality, morbidity and difficult cholecystectomy rates between two groups | patients will be followed up to the first 30 day period from discharge.
  effect of the timing on mortality, morbidity and difficult cholecystectomy in patients with acute cholecystitis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Izmir Tepecik Training and Research Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request

REFERENCES:
- [Result] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636
- [Result] Yokoe M, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Gomi H, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Kiriyama S, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF; Tokyo Guidelines Revision Committee. New diagnostic criteria and severity assessment of acute cholecystitis in revised Tokyo Guidelines. J Hepatobiliary Pancreat Sci. 2012 Sep;19(5):578-85. doi: 10.1007/s00534-012-0548-0. PMID 22872303
- [Result] Borzellino G, Sauerland S, Minicozzi AM, Verlato G, Di Pietrantonj C, de Manzoni G, Cordiano C. Laparoscopic cholecystectomy for severe acute cholecystitis. A meta-analysis of results. Surg Endosc. 2008 Jan;22(1):8-15. doi: 10.1007/s00464-007-9511-6. Epub 2007 Aug 18. PMID 17704863

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT05352087/Prot_SAP_ICF_000.pdf